CLINICAL TRIAL: NCT06850350
Title: Enhancing Veterans Long-COVID Care: A Cognitive-Sensorimotor Framework to Understand Gait and Balance Dysfunction
Brief Title: Cognitive-Sensorimotor Function in Long-COVID
Status: Not yet recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F5372-R; RX005372 (Other Grant/Funding Number: Dept Veterans Affairs)
Record Dates: First submitted 2025-02-26; First posted 2025-02-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Post-acute Sequelae of SARS-CoV-2 Infection
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Adults who previously contracted Covid-19 but do not have Long-COVID.
- Experimental: Adults who previously contracted Covid-19 and have Long-COVID.

SUMMARY:
Growing evidence indicates that many people who have chronic post-acute sequelae of SARS-CoV-2 infection (PASC) will experience ongoing neurological and musculoskeletal impairment that can affect gait and balance. Identifying the factors contributing to these impairments and how they influence functional mobility is the first step towards creating effective evaluation and treatment protocols. In this study the investigators will examine cognition, vision, proprioception, muscle strength, gait and balance in persons with and without PASC to understand how PASC may impact functional mobility through a cognitive-sensorimotor lens. Gait and balance will be studied in environments that stress cognitive and sensory abilities. Study outcomes will be critical for the development of evidence-based Veteran Health Administration diagnostic and standard-of-care protocols to address gait and balance dysfunction in Veterans with PASC for restoring their functional mobility and independence.

DETAILED DESCRIPTION:
As many as one in seven COVID-19 survivors will experience symptoms that persist more than two months after their acute illness has resolved. Growing evidence estimates that up to 30% of people who experience this chronic post-COVID disorder (aka post-acute sequelae of SARS-CoV-2 infection (PASC)) will exhibit gait and balance dysfunction. The consequences of impaired mobility are of considerable concern for the Veterans Health Administration (VHA) given that mobility is closely related to quality of life for older adults and almost half of Veterans are 65 years or older. There currently is no established VHA standard-of-care for PASC. The critical first step towards development of comprehensive clinical protocols to identify and treat PASC-related gait and balance dysfunction is understanding the contributing factors. PASC is characterized by diverse multi-organ system effects that has made it difficult to identify the causes of dysfunction. However, new data suggests frequently reported neurologic issues related to cognitive and sensorimotor impairment may be potential contributors to gait and balance dysfunction. While cognition, sensation, and muscle function can be measured in isolation, the effects of cognitive and sensory impairment on gait and balance are best detected using dual task tests (e.g., count backward by 7's while walking) that pair cognitive and motor function or tasks performed in complex environments that limit sensory feedback and/or stress sensory-motor integration (e.g., maintaining standing balance with eyes closed). However, such assessments are not included in the current recommended PASC gait and balance screening guidelines, thereby leaving a clinical gap in knowledge when evaluating and treating Veterans and non-Veterans with PASC-related gait and balance dysfunction.

Therefore, the proposed project will evaluate the effect of PASC on isolated cognitive-sensorimotor function (Aim 1), and cognitive-sensorimotor contributions to gait (Aim 2) and balance (Aim 3) dysfunction in COVID-19 survivors through an observational cross-sectional study design. Aim 1 will assess cognition, vision, proprioception, and muscle strength independent of functional task in COVID-19 survivors with and without PASC using established methods. Aim 2 will perform an instrumented assessment of gait performance of participants under a dual task scenario to stress cognition. Aim 3 will perform an instrumented assessment of postural balance under different conditions that challenge sensorimotor integration by compromising certain sensory modalities (vision, vestibular, somatosensory). A non-instrumented clinical outcome measure will also be performed as a secondary measure to evaluate a potential clinical screening tool. Based on emerging evidence, the investigators hypothesize that COVID-19 survivors with PASC will exhibit worse cognitive-sensorimotor function, dual task gait performance, and sensory-interaction balance performance than those without PASC when accounting for age, sex, and time since acute infection. PASC-induced gait and balance dysfunction has significant clinical implications as it could compromise mobility, long-term health, and quality of life of Veterans if left unaddressed.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Positive PCR or Rapid COVID-19 test in the past
* Onset of COVID-19 illness greater than 3 months prior to their participation in the study
* Self-reported ability to walk 10 meters with or without external assistance prior to COVID-19 illness

Exclusion Criteria:

* Presence of severe cardiovascular and pulmonary disease and/or neurological and musculoskeletal disorders unrelated to COVID-19 (e.g., amputation, stroke, spinal cord injury)
* Cognitive impairments precluding ability to provide informed consent.
* Severe acute COVID-19 infection requiring hospitalization or diagnosed post-intensive care syndrome.
* Presence of musculoskeletal, inflammatory, or neurological conditions mimicking Long COVID-19 symptoms (e.g., concussion within last 5 years, Chronic fibromyalgia, Myofascial pain syndrome, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who previously contracted Covid-19 and do or do not have Long-COVID.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
NIH Toolbox Cognition Battery | During single session of two hours
  The NIH Toolbox Cognition Battery to assess working memory and attention cognitive function. Working memory and attention cognitive function are quantified through performance on the List Sorting Working Memory Test and Flanker Inhibitory Control and Attention Test, respectively, administered via tablet. Raw scores from these measures can be converted to normally distributed standard (scaled) scores adjusted for age, education, sex, and/or race/ethnicity (T-Scores), as appropriate. A higher score means better performance.
Joint position sense proprioception | During single session of two hours
  Joint position sense is measured by participants' ability to accurately extend the knee joint to a target reference angle. Participants will be seated and perform nine trials where they have to replicate guided knee joint angle position of 30, 45, or 60°. The difference between guided and replicated position is recorded as the angle error, where greater error means worse proprioception.
King-Devick Test | During single session of two hours
  The King-Devick Test assesses ocular-motor function. Participants are asked to accurately and rapidly read rows of single-digit numbers displayed on a tablet. The test score is calculated as the total time required to read three test cards (each test card is approximately a full page of numbers), where faster is better.
Maximum voluntary muscle strength | During single session of two hours
  Participants will be seated and isokinetic maximum voluntary contraction is measured with a dynamometer, normalized by participant height and body mass (N-m/kg-m). Greater values mean better strength.
Dual task gait cost | During single session of two hours
  Participants will walk at their self-selected speed for 10 laps back and forth along a 10-m straight walkway with wide turns, once without a cognitive task (single task) and once with a cognitive task that stresses working memory (dual task). Difference in gait speed (m/s) is the dual task gait cost, in which higher values mean worse performance.
Modified Clinical Test of Sensory Interaction on Balance | During single session of two hours
  Participants stand on a force plate and perform four balance tasks for which participants are instructed to maintain quiet upright balance: 1) eyes open on a firm surface while focusing straight ahead (access to all three modalities), 2) eyes closed on a firm surface (compromised visual), 3) eyes open on a foam surface while focusing straight ahead (compromised somatosensory), and 4) eyes closed on a foam surface (compromised visual and somatosensory). Total CoP distance travelled (mm) of the four specific balance tasks is measured, with greater distance meaning worse performance.

SECONDARY OUTCOMES:
Mini-Balance Evaluation Systems Test | During single session of two hours
  The Mini-Balance Evaluation Systems Test is a performance-based clinical outcome measure to assess dynamic balance, including 14 items scored on a 3-level ordinal scale (total score of 28). The test assesses anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. A higher summary score means better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Major, PhD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL; Keith Edward Gordon, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No